CLINICAL TRIAL: NCT04155398
Title: A Prospective Study on the Utility of Endoscopic Ultrasound Elastography (EUS-E) for Predicting Cirrhotic-related Complications in Patients With Chronic Liver Diseases
Brief Title: EUS Elastography for Predicting Cirrhotic-related Complications
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: EUS-E study
Record Dates: First submitted 2019-11-03; First posted 2019-11-07 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Liver Fibroses
Keywords: liver stiffness; EUS elastography
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients with radiologic features suggestive of cirrhosis on abdominal imaging studies such as transabdominal ultrasound, CT or MRI and indication for variceal screening, suspected advanced liver fibrosis as detected by Fibroscan, or with clinical evidence of hypersplenism would be invited for the study
  Interventions: Procedure: EUS elastography

INTERVENTIONS:
Procedure: EUS elastography — A forward view radial echoendoscope or a forward oblique view linear echoendoscope would be used to perform focused luminal examination of varices and EUS elastography for measurement of liver stiffness and spleen stiffness.

SUMMARY:
Evaluation of the tissue stiffness as a surrogate marker of degree of liver cirrhosis has gained popularity in recent decades. Current guidelines also advocate the use of Fibroscan® machine (EchoSens, Paris, France) to detect any advanced liver fibrosis as represented by high liver stiffness, for prediction of varices development.

Apart from liver stiffness, studies have shown that spleen stiffness (SS) has been proven another useful parameter to severity of underlying portal hypertension and liver cirrhosis. However, spleen stiffness measurement by Fibroscan® is highly limited by the thickness of subcutaneous soft tissue or abdominal wall tissue, especially in obese subjects. It carries certain technical difficulty as well due to its deep-seated anatomical position.

Recently, the technique of endoscopic ultrasound elastography (EUS-E) has been described. It can overcome the limitations of Fibroscan by making measurements of liver and spleen stiffness through the gastric wall, which has a shorter distance than the abdominal wall. It also allows concomitant upper GI tract luminal examination, incorporating both esophagogastroduodenoscopy and elastography measurements into one procedure at the same time. This research study aims to prospectively study the utility of EUS-E in patients with chronic liver diseases, both in terms of diagnostic and prognostic indications for future cirrhotic-related complications.

DETAILED DESCRIPTION:
Portal hypertension is a severe consequence of chronic liver diseases and is responsible for multiple main clinical complications of liver cirrhosis. Gastroesophageal variceal bleeding is one of the notorious causes of cirrhosis-related morbidity and mortality, as a direct consequence of portal hypertension. Bleeding is usually major and carries 42% medical mortality at 6 weeks. 60% of early deaths and 40% of late deaths were attributable to bleeding. Approximately one-third of patients experienced rebleeding within 6 weeks and one-third of survivors experienced subsequent bleeds.

Assessment for portal hypertension is therefore of paramount importance. The gold standard of measurement of hepatic venous pressure gradient (HPVG) requires catheterization of the portal vein and is rarely performed in daily clinical practice due to its high invasiveness. Evaluation of the tissue stiffness as a surrogate marker of degree of liver cirrhosis has gained popularity in the recent decade. Transient elastography (TE) is one of the well proven tools to obtain liver stiffness measurements, which demonstrates good direct correlation to liver histology fibrosis staging. It also has satisfactory diagnostic performance for the prediction of clinically significant portal hypertension (HVPG > 10 mmHg) in the setting of compensated chronic liver disease or cirrhosis, with an area under receiver operating characteristics (AUROC) of 0.93. The Baveno VI criteria is one of the excellent examples to utilize TE liver stiffness measurements, all together with consideration of the platelet count, to screen out low risk patients for upper endoscopy variceal screening.

With reference to the basic anatomy, apart from liver stiffness, spleen stiffness (SS) becomes another potential quantitative parameter to the severity of underlying portal hypertension. A non-inferiority, open-label, randomized controlled trial across two hospitals in Hong Kong showed that high SS measurement by TE was independently associated with clinical significant varices. It was shown that a SSM cutoff value <41.3 kPa was sensitive and able to accurately rule out the presence of varices. Another study from Korea, with the use of acoustic radiation force impulse (ARFI) imaging, also demonstrated that SS was significantly higher in patients with varices than in those without varices (3.58 ± 0.47 vs 3.02 ± 0.49; P < 0.001). Increasing SS was observed in patients with higher grades of varices (No varix, 3.02 ± 0.49; F1, 3.39 ± 0.51; F2, 3.60 ± 0.42; F3, 3.85 ± 0.37; P < 0.001), as well as in patients who experienced variceal hemorrhage than in those who did not (3.80 ± 0.36 vs 3.20 ± 0.51; P = 0.002).

The most common way of TE is using the Fibroscan® machine (EchoSens, Paris, France). It is done by placement of a machine probe at right intercostal space over the liver parenchyma, which delivers a vibration and determines the liver stiffness by measuring the velocity of the vibration wave. It is able to measure a volume of approximately 10mm (wide) x 40mm (length) at a 25-65mm depth below the skin surface. However, it is highly limited by the thickness of subcutaneous soft tissue or abdominal wall tissue, especially in obese subjects. The spleen stiffness measurements carry certain technical difficulty as well due to its deep-seated anatomical position, particularly when it is not enlarged.

EUS elastography (EUS-E) makes use of another concept of direct tissue stiffness measurement, namely the real-time tissue elastography (RTE). It gauges the oscillation of tissue from adjacent vascular pulsation and compression, with the degree of deformation and displacement as an indicator of tissue stiffness. The tissue elasticity distribution is then represented in color superimposed on the conventional B mode image displayed. It can also be quantified in terms of Strain Ratio (SR) and Strain Histogram (SH) by machine calculation. Initially developed to differentiate benign soft tissue from malignant tumour, RTE has been used to characterize liver fibrosis in chronic liver disease of different aetiologies, as the liver is just adjacent to the stomach, which is a common scanningfield in EUS.

With such, EUS-E may offer a better option for liver and spleen stiffness measurements with the following advantages:

1. EUS is expected to have a higher success rate for LS and SS measurements, with closer distance through the gastric wall to the parenchyma. This can overcome the limitations of TE in patients with extreme body habitus, thick abdominal wall muscles and also normal spleen size.
2. Forward viewing radial echoendoscope and forward oblique viewing linear echoendoscope allow concomitant upper GI tract luminal examination, incorporating both oesophagogastroduodenoscopy (OGD) and elastography measurements into one procedure at the same time.
3. EUS can apply Doppler signals to allow detection of "deep" submucosal varices, paraesophageal and para-gastric varices that may not be routinely observed during conventional endoscopy at luminal view.

Literature search reveals utilization of other means of TE measurements, such as ARFI and 2-D shear wave elastography in SS measurements to predict clinical outcomes, such as variceal bleeding. However, there are still no relevant studies on EUS-E in terms of liver and stiffness measurements with correlation to development of cirrhotic complications, despite its more popular use and availability. Thus, investigators aim to prospectively study the utility of EUS-E in patients with chronic liver diseases, both in terms of diagnostic and prognostic indications for future cirrhotic-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with radiologic features suggestive of cirrhosis on abdominal imaging studies such as transabdominal ultrasound, CT or MRI and indication for variceal screening
* Patients with suspected advanced liver fibrosis as detected by Fibroscan
* Patients with clinical evidence of hypersplenism
* Age > 18 years
* Written informed consent available

Exclusion Criteria:

* Patients with features of decompensated cirrhosis, such as history of ascites, prior variceal bleeding, hepatic encephalopathy, hepatorenal syndrome
* Patients with history of hepatocellular carcinoma
* Patients with history of liver transplant or TIPS or shunting surgery
* Patients with portal and/or mesenteric vein thrombosis
* Moribund patients from terminal illnesses
* Patients with terminal malignancy
* Contraindications for endoscopy
* Unable to provide written informed consent
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with radiologic features suggestive of cirrhosis on abdominal imaging studies such as transabdominal ultrasound, CT or MRI and indication for variceal screening, suspected advanced liver fibrosis as detected by Fibroscan, or with clinical evidence of hypersplenism would be invited for the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Inter-observer and intra-observer variability of liver and spleen stiffness measurements by EUS-E among endoscopists with different EUS experience | peri-procedure
  Inter-observer and intra-observer variability of liver and spleen stiffness measurements by EUS-E among endoscopists with different EUS experience
Diagnostic performance of liver and spleen stiffness measurements by EUS-E to predict variceal development and/or bleeding | Follow up for 2 years after index study endoscopy
  Diagnostic performance of liver and spleen stiffness measurements by EUS-E to predict variceal development and/or bleeding

SECONDARY OUTCOMES:
Diagnostic performance of liver and spleen stiffness measurements by EUS-E to predict other liver cirrhosis complications (eg, ascites, hepatic encelopathy, etc) | Follow up for 2 years after index study endoscopy
  Diagnostic performance of liver and spleen stiffness measurements by EUS-E to predict other liver cirrhosis complications (eg, ascites, hepatic encelopathy, etc)
Correlation of liver fibrosis by EUS-E to Fibroscan | Follow up for 2 years after index study endoscopy
  Correlation of liver fibrosis by EUS-E to Fibroscan
Adverse events related to procedure | peri-procedure
  Adverse events related to procedure

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tang, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No